CLINICAL TRIAL: NCT05009407
Title: CD160 Ans Corneal Graft: Expression in Corneal Vessels
Brief Title: CD160 Expression in Corneal Vessels
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO21062
Record Dates: First submitted 2021-08-03; First posted 2021-08-17 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Corneal Graft Rejection; CD160; Angiogenesis; Lymphangiogenesis
Keywords: Corneal Graft Rejection; CD160; Angiogenesis; lymphangiogenesis
MeSH Terms: interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HOSTS: patients ongoing corneal transplantation procedure which a full-thickness cornea from the host is replaced by a graft from a donor
  Interventions: Biological: Immunohistochemistry and clinical analyses on patients and corneas
- DONORS: grafts from donors that would be analyzed
  Interventions: Biological: Immunohistochemistry and clinical analyses on patients and corneas

INTERVENTIONS:
Biological: Immunohistochemistry and clinical analyses on patients and corneas — Immunohistochemistry and clinical analyses on patients and corneas

SUMMARY:
Despite improvements in corneal transplantation, anti-angiogenic and anti-lymphangiogenic factors remain to be be identified. CD160 is an anti-angiogenic target: its expression seems to be restricted to some immune cells and to activated endothelial cells. We hypothesized that CD160 is expressed in blood and lymphatic human corneal neovessels and is involved in corneal graft rejection pathogenesis

DETAILED DESCRIPTION:
After informed consent, patients enrolled for corneal graft surgery at the Robert Debré University Hospital, Reims, France, will be included.

Routine general and eye examination including cornea photographs will be performed.

During surgery, a quarter of patients' cornea and of donors' corneoscleral rim will be spared for immunohistochemistry analyzes.

ELIGIBILITY:
inclusion criteria :

* 18-year-old or more patients
* enrolled for penetrating keratoplasty or deep anterior lamellar keratoplasty surgeries at the Robert Debré University Hospital, Reims, France
* considered able to give an informed written consent exclusion criteria :
* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-year-old or more patients enrolled for penetrating keratoplasty or deep anterior lamellar keratoplasty surgeries at the Robert Debré University Hospital, Reims, France
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-07-21 (Estimated); Study Completion 2024-07-21 (Estimated)

PRIMARY OUTCOMES:
Micro-vascular densities | 1 year
  neovascularization scores quantification of blood (anti-ERG+/anti-D2-40-) and lymphatic (anti-ERG+/anti-D2-40+) vascular structures ; Percentages of those vascular structures marked with anti-CD160

SECONDARY OUTCOMES:
Percentages of those vascular structures marked with anti-CD160 and/or CD105 and/or aSMA | 1 year
Evaluation of clinical blood vascular densities on photographs with help of ImageJ software | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France